CLINICAL TRIAL: NCT05438043
Title: A Phase 3b, Multicenter, Open-label, Daratumumab Long-term Extension Study
Brief Title: A Study of Daratumumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109200; 54767414MMY3030 (Other: Janssen Research & Development, LLC); 2021-006494-33 (EudraCT Number); 2022-500138-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; carfilzomib; Dexamethasone; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Participants will receive a single dose of daratumumab 16 milligrams per kilograms (mg/kg) intravenous (IV) or 1800 mg subcutaneous (SC) infusion on Cycle 1 Day 1 (28-day cycle), as monotherapy or in combination with standards of care treatment (that is, pomalidomide and dexamethasone, lenalidomide and dexamethasone, carfilzomib and dexamethasone) or standards of care treatment alone, depending on the treatment received in the parent study. Participants who received daratumumab IV during the parent study, will have an option to switch to daratumumab SC on Day 1 of any cycle during this long-term extension study.
  Interventions: Drug: Daratumumab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Pomalidomide

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered either intravenously or subcutaneously.
  Other Names: JNJ-54767414
Drug: Carfilzomib — Carfilzomib will be administered intravenously.
Drug: Dexamethasone — Dexamethasone will be administered either orally or intravenously.
Drug: Lenalidomide — Lenalidomide will be administered orally.
Drug: Pomalidomide — Pomalidomide will be administered orally.

SUMMARY:
The purpose of this study is to provide ongoing access to study treatments for participants with multiple myeloma or smoldering multiple myeloma benefiting from treatment in certain Janssen Research and Development (R&D) studies that use daratumumab as part of the study treatment regimen: access for all participants regardless of treatment group in daratumumab studies and access to participants in daratumumab-containing arms in the non-daratumumab studies will be allowed from studies which have reached clinical cutoff for final analysis. Certain long-term safety data will continue to be collected from study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be actively receiving daratumumab (either as monotherapy or in combination with other study treatment) in certain Janssen research and development (R&D) studies or receiving other study treatment in a Janssen R&D daratumumab study for participants with multiple myeloma or smoldering multiple myeloma which has reached clinical cutoff for final analysis continue to benefit from study treatment, not have experienced disease progression or unmanageable toxicity while receiving daratumumab, not have met the withdrawal criteria set forth in the parent study, and have had the last dose of study treatment within the previous 3 months
* Investigator's assessment that the benefit of continued study treatment will outweigh the risks
* A female participant of childbearing potential must have a negative pregnancy test at screening and must agree to further serum or urine pregnancy tests during the study
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 3 months after receiving the last dose of study treatment
* Must sign an informed consent form (ICF; or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Has taken any disallowed therapies or treatment for the disease under study between the completion of the parent study and the planned first dose of study treatment
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Known allergies, hypersensitivity, or intolerance to study treatments or their excipients (refer to the daratumumab investigator brochure (IB) and local country prescribing information for dexamethasone, carfilzomib, pomalidomide, and lenalidomide)
* Vaccinated with an investigational vaccine (except for Coronavirus disease [COVID-19])or live attenuated or replicating viral vector vaccines within 4 weeks prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | 3 years 7 months
  Number of participants with SAEs will be reported. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product.
Number of Participants with AEs of Special Interest (AESI) | 3 years 7 months
  Number of participants with AESI, that is, reactivation of HBV infection, will be reported.
Number of Participants with Pregnancies or Partner Pregnancies | 3 years 7 months
  Number of participants with pregnancies or partner pregnancies will be reported using the appropriate pregnancy notification form.
Number of Participants with Abnormal Pregnancies as SAE | 3 years 7 months
  Number of Participants with Abnormal Pregnancies as SAE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (85):
- United States (7):
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barnes-jewish Hospital, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai - The Derald H. Ruttenberg, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Baylor University Medical Center, Dallas, Texas
- ZNA Stuivenberg, Antwerp, Belgium
- Brazil (3):
  - Liga Norte Riograndense Contra O Cancer, Natal
  - COI Clinicas Oncologicas Integradas, Rio de Janeiro
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
- China (19):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Chaoyang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - West China Hospital Si Chuan University, Chengdu
  - Fujian Medical University, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - First Affiliated Hospital Medical School of Zhejiang University, Hangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin cancer hospital, Tianjin
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Henan Cancer Hospital, Zhengzhou
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Všeobecná fakultní nemocnice v, Prague
- Aarhus University Hospital, Aarhus N, Denmark
- France (4):
  - Centre Hospitalier Universitaire (CHU) de Caen, Caen
  - CHU Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Haut Leveque, Pessac
- Germany (3):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
- Greece (2):
  - Alexandra General Hospital of Athens, Athens Attica
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
- Italy (2):
  - Universita Degli Studi di Roma Tor Vergata, Roma
  - Sapienza University of Rome, Roma
- Poland (2):
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
- Russia (8):
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Republican Hospital named by V.A.Baranova, Petrozavodsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - City Hospital No.15, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Oncology Dispensary of Komi Republic, Syktyvkar
- South Korea (7):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (17):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Del Mar, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hosp. Gral. Univ. J.M. Morales Meseguer, Murcia
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Univ. Dr. Peset, Valencia
- Ege Universitesi Tip Fakultesi, Izmir, Turkey (Türkiye)
- Ukraine (4):
  - CNE Clinical Center of Oncology Hematology Transplantology and Palliative Care of the Cherkasy RC, Cherkasy
  - Municipal Non-Commercial Enterprise City Clinical Hospital No 4 of Dnipro City Council, Dnipro
  - MNE Regional Oncology Center, Kharkiv
  - Vinnytsya Regional Clinical Hospital named after M.I.Pirogov, Vinnitsa
- United Kingdom (2):
  - St James University Hospital, Leeds
  - Royal Marsden Hospital, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency